CLINICAL TRIAL: NCT00337246
Title: A Randomized Phase II Trial of Fludarabine, Cyclophosphamide and Mitoxantrone (FCM) With or Without Rituximab in Previously Treated Chronic Lymphocytic Leukemia
Brief Title: Combination Chemotherapy With or Without Rituximab in Treating Patients With Previously Treated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CTRU-NCRI-UKCLL01-FCM/FCM-R; CDR0000485181 (Registry Identifier: PDQ (Physician Data Query)); EU-20626; ROCHE-NCRI-UKCLL01-FCM/FCM-R; ISRCTN77546448; EUDRACT-2004-003982-34
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-05

CONDITIONS: Leukemia
Keywords: refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; fludarabine phosphate; Mitoxantrone

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, cyclophosphamide, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving combination chemotherapy together with rituximab may kill more cancer cells. It is not yet known whether giving combination chemotherapy together with rituximab is more effective than combination chemotherapy alone in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase II trial is studying how well giving combination chemotherapy with or without rituximab works in treating patients with previously treated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the efficacy and safety of fludarabine, cyclophosphamide, and mitoxantrone hydrochloride with or without rituximab in patients with previously treated chronic lymphocytic leukemia.
* Determine the overall response rate, defined as complete or partial remission, in these patients.

Secondary

* Determine the proportion of patients with undetectable minimal residual disease.
* Determine the 2-year progression-free survival of these patients.
* Determine the 2-year overall survival of these patients.
* Determine the toxicity of this regimen.

OUTLINE: This is a randomized, controlled, open-label, parallel group, multicenter study. Patients are stratified according to prior treatment with fludarabine (refractory vs not refractory or naive). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral fludarabine* and oral cyclophosphamide* on days 1-5 and mitoxantrone hydrochloride IV on day 1.
* Arm II: Patients receive fludarabine*, cyclophosphamide*, and mitoxantrone hydrochloride as in arm I. Patients also receive rituximab IV on day 1.

NOTE: *If the oral regimen is not tolerated, patients may receive fludarabine IV and cyclophosphamide IV on days 1-3.

Treatment in both arms repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 3 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia requiring therapy
* Previously treated with ≥ 1 chemotherapeutic regimen

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 12 weeks
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective contraception for 4 weeks before, during, and for 6 months after completion of study treatment
* Fertile male patients must use effective contraception during and for 6 months after completion of study treatment
* No history of anaphylaxis after exposure to rat or mouse-derived complementary-determining region (CDR)-grafted humanized monoclonal antibodies
* No toxicity attributable to purine analogues (e.g., autoimmune hemolytic anemia, neurological toxicity, or allergy)
* No active infection
* No other severe (particularly cardiac or pulmonary) diseases or mental disorders that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior fludarabine (or other purine analogues) combined with cyclophosphamide and mitoxantrone hydrochloride
* No prior rituximab, either alone or in combination with chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2005-07; Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate as measured by NCI Response Criteria

SECONDARY OUTCOMES:
Proportion of patients with undetectable minimal residual disease
Progression-free survival at 2 years
Overall survival at 2 years
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillmen, MD, Study Chair — Leeds General Infirmary
Locations (16):
- United Kingdom (16):
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St Helier Hospital, Carshalton, England
  - Darent Valley Hospital, Dartford Kent, England
  - Medway Maritime Hospital, Gillingham Kent, England
  - Leeds General Infirmary at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals NHS Trust, Liverpool, England
  - Maidstone Hospital, Maidstone, England
  - Christie Hospital NHS Trust, Manchester, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - Kent and Sussex Hospital, Tunbridge Wells, Kent, England
  - Wishaw General Hospital, Wishaw, England
  - Monklands General Hospital, Airdrie, Scotland
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Result] Hillmen P, Cohen DR, Cocks K, Pettitt A, Sayala HA, Rawstron AC, Kennedy DB, Fegan C, Milligan DW, Radford J, Mercieca J, Dearden C, Ezekwisili R, Smith AF, Brown J, Booth GA, Varghese AM, Pocock C; NCRI CLL Sub-Group. A randomized phase II trial of fludarabine, cyclophosphamide and mitoxantrone (FCM) with or without rituximab in previously treated chronic lymphocytic leukaemia. Br J Haematol. 2011 Mar;152(5):570-8. doi: 10.1111/j.1365-2141.2010.08317.x. Epub 2011 Jan 14. PMID 21231927